CLINICAL TRIAL: NCT04507620
Title: Effect of Cervical Neck Collar and Head Blocks Strapped on the Backboard on Optic Nerve Sheath Diameter
Brief Title: Effect of Cervical Immobilization on Optic Nerve Sheath Diameter
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Elbahnasawy, MD, consultant of emergency medicine and traumatology, Tanta University
Other Study IDs: 33935/7/20
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Optic Nerve Sheath Diameter; Point of Care Ultrasound
Keywords: cervical immobilization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cervical neck collar
  Interventions: Device: cervical neck collar
- head blocks strapped on the backboard
  Interventions: Device: cervical neck collar

INTERVENTIONS:
Device: cervical neck collar — devices used for cervical immobilization
  Other Names: head blocks strapped on the backboard

SUMMARY:
Effect of Cervical Immobilization on Optic Nerve Sheath Diameter

DETAILED DESCRIPTION:
Two cervical immobilization devices will be used in this study named cervical neck collar and head blocks strapped on the backboard and optic nerve diameter will be measured using point of care ultrasound and compare the effect of each type of cervical immobilisation on optic nerve sheath diameter.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers aged more than 18 years

Exclusion Criteria:

* Hx of stroke

  * Inability to consent,
  * Inability to lay flat on a bed or table for 15 min in duration,
  * History of glaucoma, globe injury, lens implant,
  * Recent refractive surgery (within the past 60 days).
  * Uncontrolled hypertension

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This prospective study will be done on 100 medical students, emergency medicine and traumatology residents and assistant lecturers ,Tanta university faculty of medicine, healthy volunteers during a period of 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Effect of cervical neck collar and head blocks strapped on the backboard on Optic Nerve Sheath Diameter | 6 month
  effect of cervical neck collar and head blocks strapped on the backboard on optic nerve sheath diameter, measured by point of care ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Elbahnasawy, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No